CLINICAL TRIAL: NCT07071610
Title: A Phase II, Randomized, Double-Blind, Vehicle-Controlled Study to Evaluate the Efficacy and Safety of LNK01004 Ointment in Adults With Atopic Dermatitis
Brief Title: A Study to Evaluate the Efficacy and Safety of LNK01004 Ointment in Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lynk Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LK004201
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vehicle (Placebo Comparator): Participants applied vehicle ointment BID for 8 weeks in DB period.
  Interventions: Drug: Vehicle
- LNK01004 ointment 0.3% (Experimental): Participants applied LNK01004 ointment 0.3% BID for 8 weeks in DB period.
  Interventions: Drug: LNK01004 ointment 0.3%
- LNK01004 ointment 1.0% (Experimental): Participants applied LNK01004 ointment 1.0% BID for 8 weeks in DB period.
  Interventions: Drug: LNK01004 ointment 1.0%

INTERVENTIONS:
Drug: LNK01004 ointment 0.3% — LNK01004 ointment 0.3% BID
  Arms: LNK01004 ointment 0.3%
Drug: LNK01004 ointment 1.0% — LNK01004 ointment 1.0% BID
  Arms: LNK01004 ointment 1.0%
Drug: Vehicle — vehicle BID
  Arms: Vehicle

SUMMARY:
This study will evaluate the efficacy and safety of two concentrations (0.3 percent [%] and 1%) of twice daily LNK01004 ointment for the topical treatment in adult subjects with atopic dermatitis. This is a multicenter, randomized, double-blind, vehicle-controlled, 3-arm, parallel-group, dose-finding study in adult subjects with atopic dermatitis. Two concentrations of LNK01004 ointment (0.3% and 1%) and a vehicle control ointment will be equally randomized and evaluated following application to all atopic dermatitis lesions (except on the scalp) twice daily (morning and evening) for 8 weeks.

This study will consist of 3 periods: up to 4 weeks screening, 8 weeks double-blind treatment, and 2 weeks post-treatment follow-up.

Approximately 75 subjects (25 subjects for each group) with moderate to severe AD will be enrolled overall.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years at screening.
* Diagnosis of AD as defined by the Hanifin and Rajka (1980) criteria for at least 3 months at screening.
* Stable course of AD (not spontaneously improving or rapidly deteriorating) as determined by the investigator in the 3 weeks before screening.
* IGA score of 3 to 4 at screening and baseline.
* BSA of AD involvement, excluding the Scalp, Palms, and Soles, of 5% to 35% at screening and baseline.
* Willingness to avoid pregnancy or fathering children based on the criteria as outlined in the protocol.

Exclusion Criteria:

* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would pose a significant risk to the participant or interfere with the interpretation of study data.
* Concurrent conditions and history of:

  * Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before Baseline.
  * Active acute bacterial, fungal, or viral skin infection within 1 week before Baseline.
  * Any other concomitant skin disorder, pigmentation, or extensive scarring that, in the opinion of the investigator, may interfere with the evaluation of AD lesion.
  * Any other concomitant non-skin disorder with the treatment that may interfere with the evaluation of AD.
* Use of any of the following treatments within the indicated period before Baseline:

  * 6 weeks: Dupilumab
  * 5 half-lives or 12 weeks, whichever is longer: biologic agents (except dupilumab).
  * 4 weeks: Janus kinase (JAK) inhibitors.
  * 5 half-lives or 4 weeks, whichever is longer: Systemic therapy for AD, including but not limited to corticosteroids, methotrexate, cyclosporine, azathioprine, phosphodiesterase type 4 (PDE4)-inhibitors, Ultraviolet (UV) light therapy, or traditional Chinese medicine.
  * 2 weeks: Sedating antihistamines.
  * 1 week: Topical AD treatments (except topical emollient treatments), including but not limited to TCS, TCIs, or topical PDE-4 inhibitors.
* Hepatitis B surface antigen (HBs Ag) positive (+); HCV ribonucleic acid (RNA) detectable in any subject with anti-HCV antibody (HCV Ab); Human immunodeficiency virus (HIV) positive (+).
* Participants with the following hematologic abnormalities at screening:

  * ALT or AST ≥ 2 × ULN
  * TBiL ≥ 2 × ULN
  * Creatinine ≥ 1.5 × ULN
* History of alcoholism or drug addiction within 6 months before screening or current alcohol or drug use.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before Baseline with another investigational medication or current enrollment in another investigational drug protocol.
* Participants who are pregnant, nursing, or planning a pregnancy during the study period.
* Participants with known allergies to components or excipients of the test drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Mean Percentage Change From Baseline in Eczema Area and Severity Index (EASI) Score at Week 8 | Baseline to week 8
  EASI is a validated composite scoring system integrating the proportion of the body region (area) involved and the intensity of key signs of atopic dermatitis (AD). The EASI score examines 4 regions of the body and weights them for participants 8 years of age and older as follows: Head/Neck (H) = 0.1, Upper limbs (UL) = 0.2, Trunk (T) = 0.3, and Lower limbs (LL) = 0.4. Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement). The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The total EASI score ranges from 0 to 72. A higher score indicated worse disease status, and a negative change from baseline indicated improvement.

SECONDARY OUTCOMES:
Change From Baseline in Eczema Area and Severity Index (EASI) Score at Week 8 | Baseline to week 8
  EASI is a validated composite scoring system integrating the proportion of the body region (area) involved and the intensity of key signs of atopic dermatitis (AD). The EASI score examines 4 regions of the body and weights them for participants 8 years of age and older as follows: Head/Neck (H) = 0.1, Upper limbs (UL) = 0.2, Trunk (T) = 0.3, and Lower limbs (LL) = 0.4. Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement). The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The total EASI score ranges from 0 to 72. A higher score indicated worse disease status, and a negative change from baseline indicated improvement.
Percentage of Participants Who Achieve a ≥ 75% Improvement From Baseline in EASI (EASI-75) at Week 8 | Baseline to week 8
  EASI is a validated composite scoring system integrating the proportion of the body region (area) involved and the intensity of key signs of atopic dermatitis (AD). The EASI score examines 4 regions of the body and weights them for participants 8 years of age and older as follows: Head/Neck (H) = 0.1, Upper limbs (UL) = 0.2, Trunk (T) = 0.3, and Lower limbs (LL) = 0.4. Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement). The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The total EASI score ranges from 0 to 72. A higher score indicated worse disease status, and a negative change from baseline indicated improvement.
Percentage of Participants Who Achieve a ≥ 90% Improvement From Baseline in EASI (EASI-90) at Week 8 | Baseline to week 8
  EASI is a validated composite scoring system integrating the proportion of the body region (area) involved and the intensity of key signs of atopic dermatitis (AD). The EASI score examines 4 regions of the body and weights them for participants 8 years of age and older as follows: Head/Neck (H) = 0.1, Upper limbs (UL) = 0.2, Trunk (T) = 0.3, and Lower limbs (LL) = 0.4. Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement). The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The total EASI score ranges from 0 to 72. A higher score indicated worse disease status, and a negative change from baseline indicated improvement.
Percentage of Participants Who Achieve a ≥ 50% Improvement From Baseline in EASI (EASI-50) at Week 2 | Baseline to week 2
  EASI is a validated composite scoring system integrating the proportion of the body region (area) involved and the intensity of key signs of atopic dermatitis (AD). The EASI score examines 4 regions of the body and weights them for participants 8 years of age and older as follows: Head/Neck (H) = 0.1, Upper limbs (UL) = 0.2, Trunk (T) = 0.3, and Lower limbs (LL) = 0.4. Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement). The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The total EASI score ranges from 0 to 72. A higher score indicated worse disease status, and a negative change from baseline indicated improvement.
Percentage of Participants Achieving an Investigator's Global Assessment (IGA) Score of 0 to 1 Who Have an Improvement of ≥ 2 Points at Week 8 | Baseline to week 8
  IGA is an assessment scale used to determine severity of atopic dermatitis (AD) and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). An IGA responder was defined as a participant achieving an IGA score of 0 to 1 and an IGA score improvement at least 2 from baseline.
Percentage of Participants Achieving ≥4-Point Improvement in WI-NRS Pruritus Score at Week 8 | Baseline to week 8
  The number of participants achieving a ≥4-point improvement from Baseline in WI-NRS score is presented. The WI-NRS is a simple, single item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the subject experienced in the previous 24 hours. Higher scores indicate greater symptom severity.
Number of Participants with Any Treatment-emergent Adverse Event (TEAE) | Baseline to week 10
  An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug-related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. TEAEs were defined as any AEs with an onset date during or after the first study treatment dose.
Plasma Concentration of LNK01004 | week 4,week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
This is due to proprietary and regulatory considerations. The data will remain confidential to protect intellectual property and participant privacy.